CLINICAL TRIAL: NCT06219733
Title: A Phase II, Open-Label, Randomized, Controlled Study to Evaluate Efficacy and Safety of Vactosertib and Imatinib Combination in Patients with Advanced Desmoid Tumor (Aggressive Fibromatosis) Compared with Imatinib Monotherapy
Brief Title: Vactosertib and Imatinib Combination in Patients with Advanced Desmoid Tumor/aggressive Fibromatosis (DT/AF)
Acronym: MP-VAC-206
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Changing trial strategy
Sponsor: MedPacto, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP-VAC-206
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Dermoid
MeSH Terms: conditions — Dermoid Cyst | interventions — vactosertib; Imatinib Mesylate

STUDY DESIGN:
Intervention Model Description: 1:1 allocation into two arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vactosertib and imatinib combination (Experimental): Vactosertib 200 mg PO BID 5 days on / 2 days off in combination with imatinib 400 mg PO QD daily
  Interventions: Drug: Vactosertib
- Imatinib alone (Active Comparator): Imatinib 400 mg PO QD daily
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Vactosertib — 200 mg PO BID 5 days on / 2 days off
  Arms: Vactosertib and imatinib combination
Drug: Imatinib — Imatinib 400 mg PO QD daily
  Arms: Imatinib alone

SUMMARY:
Vactosertib and imatinib combination in patients with advanced desmoid tumor/aggressive fibromatosis (DT/AF) compared with imatinib monotherapy

DETAILED DESCRIPTION:
This is an open-label, multi-center, randomized controlled study to evaluate the safety and efficacy of vactosertib 200 mg BID in combination with imatinib versus imatinib alone.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Be capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Provision of signed and dated, written informed consent form prior to any mandatory study specific procedures, sampling, and analyses.
3. Have diagnosed with DT/AF histologically.
4. Meet one of the following criteria to be eligible:

   1. Progression by radiographic image by RECIST v1.1 or increase in tumor size equal to, or greater than (≥) 10% within 6 months prior to C1D1
   2. Patients with documented symptomatic disease related to DT/AF including pain, limitation of function, etc.
5. Have at least one measurable lesion based on RECIST v1.1: Target lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
6. Have a performance status of ≤ 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status.
7. Be able to swallow tablets and absorb vactosertib and imatinib.
8. Have adequate organ function as indicated by the following laboratory values
9. Have no history of additional malignancy that is progressing or has required active treatment within the past 3 years, with the exception of basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, or in situ cervical cancer, or have undergone potentially curative therapy with no evidence of that disease recurrence.
10. Be able to provide a newly acquired (within 6 months prior to C1D1) tumor sample during screening (preferred) or provide an available archived tumor sample. At least 10 subjects in each treatment group should be able to provide newly acquired (within 6 months prior to C1D1) tumor sample. Tumor lesions used for newly acquired biopsies should not be target lesions, unless there are no other lesions suitable for biopsy, and in this instance only core needle (not excisional/incisional) biopsy is allowed. Samples with limited tumor content and fine needle aspirate specimens are not acceptable. The tumor specimen should be of sufficient quantity to allow for exploratory biomarker analyses and is preferred in formalin fixed paraffin embedded blocks.
11. For a female of childbearing potential, have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required (Refer to Section 4.6.2).
12. For a female of childbearing potential, be willing to use an adequate method of contraception as outlined in the protocol for the course of the study through 90 days after the last dose of study treatment.
13. For a male subject with a female partner(s) of child-bearing potential, must agree to use an adequate method of contraception as outlined in the protocol, starting with the first dose of study therapy through 90 days after the last dose of study therapy. Males with pregnant partners must agree to use an adequate method according to the protocol (Refer to Section 4.6.2) no additional method of contraception is required for the pregnant partner.

Exclusion Criteria:

1. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

   Note: Subjects who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
2. Has exposed to vactosertib or imatinib for treatment purpose
3. Before the first dose of trial treatment (<2 weeks prior to first dose):

   1. Has received prior systemic cytotoxic chemotherapy
   2. Has received antineoplastic biological therapy
   3. Had major surgery *Note: Subjects should recover from therapy related toxicity to less than CTCAE Grade 2 in order to participate in this trial.
4. Is taking prohibited medications when using vactosertib as following (Refer to Appendix D Prohibited Concurrent Medications with Vactosertib (Ver 06Mar2020)
5. A minimal washout period of 5 half-lives for the following drugs is mandatory prior to the first dosing.

   1. Concurrent use of drugs or foods that are known strong CYP3A4 inhibitors including but not limited to grapefruit juice, itraconazole, ketoconazole, lopinavir/ritonavir, mibefradil, voriconazole. The topical use of these medications (if applicable), such as 2% ketoconazole cream, may be allowed.
   2. Concurrent use of drugs that are known potent CYP3A4 inducers including but not limited to phenytoin, rifampin, St. John's wort.
   3. Concurrent use of drugs that are CYP3A4, CYP1A2, CYP2B6 substrates with narrow therapeutic indices including but not limited to theophylline, astemizole, cisapride, cyclosporine, dihydroergotamine, ergotamine, sirolimus, tacrolimus, terfenadine (astemizole, cisapride, and terfenadine have been withdrawn from the US market).
   4. Concurrent use of drugs that are sensitive CYP3A4, CYP1A2, CYP2B6 substrates including but not limited to efavirenz, darunavir, dasatinib, everolimus, lopinavir, midazolam, sirolimus, ticagrelor.
6. Has severe hypersensitivity to vactosertib, imatinib, and/or any of its excipients
7. Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
8. Has an active infection requiring systemic therapy. Has a known history of Hepatitis B (defined as HBsAg reactive) or known active Hepatitis C virus (defined as HCV RNA is detected) infection.
9. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association Class III/IV), uncontrolled hypertension (≥150/90mmHg), unstable angina pectoris or myocardial infarction (≤6 months prior to screening), uncontrolled cardiac arrhythmia, clinically significant cardiac valvulopathy requiting treatment, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the subject to give written informed consent.
10. QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥450 ms in male and ≥470 ms in female calculated from 12-lead ECGs.
11. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.
12. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study.
13. Has been unable to comply with study procedures (including, but not limited to, the completion of patient report outcomes (PROs) or the PRO questionnaires are not available in the subject's preferred language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
progression-free survival | 28 days
  To evaluate the progression-free survival (PFS) of vactosertib and imatinib combination compared with imatinib alone up to 2 years. The subject will be assessed until disease progression is observed or death, which comes first. The disease progression will be assessed using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 Criteria. The date of progression will be determined by a blinded, independent, central radiologic review (BICR).

CONTACTS AND LOCATIONS:
Overall Officials: Sunjin Hwang, MD, Study Director — MedPacto, Inc.
Locations (1):
- Yeonsei University Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No